CLINICAL TRIAL: NCT03304483
Title: Cardiovascular Effects of Ultramarathon Running
Brief Title: Cardiovascular Responses to Spartathlon Running
Acronym: Spartathlon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Cardiologist, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 84542
Record Dates: First submitted 2017-09-28; First posted 2017-10-09 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Disorder Heart
MeSH Terms: conditions — Heart Diseases | interventions — Running

STUDY DESIGN:
Intervention Model Description: athletes participating in the ultra marathon running
Masking Description: Before and after the race
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes (Experimental): 246-km running
  Interventions: Other: 246-km running

INTERVENTIONS:
Other: 246-km running — Spartathlon 2017

SUMMARY:
The aim of this study is to examine the cardiovascular effects of ultramarathon running and their relation to performance.

DETAILED DESCRIPTION:
The purpose of the study is to determine the changes of cardiovascular morphology and function after an ultramarathon race. 50 entrants to the "Spartathlon 2017" 246-km running race will participate in the study. Cardiac and arterial morphology and function tests will be conducted one day before the race and within 20 minutes of race completion.

ELIGIBILITY:
Inclusion Criteria:

* Runners at least 18 years old, healthy and sufficiently trained.
* Runners being accepted to participate in the Spartathlon race according to the eligibility criteria (http://www.spartathlon.gr/en/registration-en.html)
* Runners who will volunteer to be examined pre- and post the race

Exclusion Criteria:

* Runners with chronic diseases
* Runners receiving any medication

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change of right ventricular function after one day ultra-marathon running | before and after 1 day running
  Echocardiographic study of left ventricular function

SECONDARY OUTCOMES:
Change of left ventricular function after one day ultra-marathon running | before and after 1 day running
  Echocardiographic study of left ventricular function
Change of carotid artery function after one day ultra-marathon running | before and after 1 day running
  Echocardiographic study of carotid arteries

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Kouidi, Professor, Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Laboratory of Sports Medicine, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
No personal details will be shared. Only the results of the measurements will be available

REFERENCES:
- [Background] Seedhouse EL, Walsh ML, Blaber AP. Heart rate, mean arterial blood pressure, and pulmonary function changes associated with an ultraendurance triathlon. Wilderness Environ Med. 2006 Winter;17(4):240-5. doi: 10.1580/pr27-05-r1.1. PMID 17219787
- [Background] Millet GP, Millet GY. Ultramarathon is an outstanding model for the study of adaptive responses to extreme load and stress. BMC Med. 2012 Jul 19;10:77. doi: 10.1186/1741-7015-10-77. PMID 22812424
- [Background] Cote AT, Phillips AA, Foulds HJ, Charlesworth SA, Bredin SS, Burr JF, Koehle MS, Warburton DE. Sex differences in cardiac function after prolonged strenuous exercise. Clin J Sport Med. 2015 May;25(3):276-83. doi: 10.1097/JSM.0000000000000130. PMID 25010150
- [Background] Jee H, Park J, Oh JG, Lee YH, Shin KA, Kim YJ. Effect of a prolonged endurance marathon on vascular endothelial and inflammation markers in runners with exercise-induced hypertension. Am J Phys Med Rehabil. 2013 Jun;92(6):513-22. doi: 10.1097/PHM.0b013e31829232db. PMID 23685440
- [Result] Blaber AP, Walsh ML, Carter JB, Seedhouse EL, Walker VE. Cardiopulmonary physiology and responses of ultramarathon athletes to prolonged exercise. Can J Appl Physiol. 2004 Oct;29(5):544-63. doi: 10.1139/h04-035. PMID 15507692